CLINICAL TRIAL: NCT04750395
Title: Open-label Randomized Controlled Trial of Oral Transmucosal Haloperidol and Olanzapine in the Treatment of Terminal Delirium
Brief Title: Comparing Haloperidol and Olanzapine in Treating Terminal Delirium
Acronym: HALOLAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HCA Hospice Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-HALOLAN
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Delirium; Terminal Illness
Keywords: Haloperidol; Olanzapine; terminal delirium; home hospice
MeSH Terms: conditions — Delirium | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, randomized controlled trial. Patients will be randomly assigned to one of two groups as part of follow-up management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haloperidol (Experimental): Every 24 hours, patients will receive two regular doses of OT Haloperidol 2.5mg. Patients may also receive up to two breakthrough doses within a minimum interval of one hour from the last dose. In total, up to four doses of medication will be prepared.
  Interventions: Drug: Haloperidol Solution
- Olanzapine (Experimental): Every 24 hours, patients will receive two regular doses of OT Olanzapine 5.0mg. Patients may also receive up to two breakthrough doses within a minimum interval of one hour from the last dose. In total, up to four doses of medication will be prepared.
  Interventions: Drug: Olanzapine Tablets

INTERVENTIONS:
Drug: Haloperidol Solution — Oral transmucosal haloperidol solution 2.5mg
  Arms: Haloperidol
Drug: Olanzapine Tablets — Oral transmucosal olanzapine tablet 5.0mg
  Arms: Olanzapine

SUMMARY:
As patients with terminal illness enter the dying phase, they may experience symptoms of restlessness, agitation, or cognitive disturbance, known as terminal delirium. In community care, pharmacological therapies are utilized to manage the syndrome, the most commonly used being neuroleptics haloperidol and olanzapine.

However, there is currently a dearth of studies on the efficacy and safety between haloperidol and olanzapine in the community palliative care setting; existing studies involve non-terminal patients in the hospital suffering from acute delirium. To fill this gap, an open-label randomized clinical trial is proposed to compare the effects of haloperidol and olanzapine in the management of terminal delirium in home hospice patients who are imminently dying. Key outcome measures are the reduction of delirium symptoms and the reduction of agitation. Secondary outcome is comparing the adverse effect burden on patients.

DETAILED DESCRIPTION:
Our study defines "terminal delirium" as an episode of delirium that occurs during the dying phase, usually 72 hours before death. Episodes of delirium in the dying phase may be described as "terminal restlessness" or "terminal delirium". The use of the label "terminal" implies a causal relationship between the dying phase and the delirium, although the aetiology is often multi-factorial.

A prospective, open-label, randomized controlled trial was designed. When a home hospice clinician identifies a patient who meets inclusion criteria, their proxy (i.e. family caregivers) will be approached by the study team and invited to participate in the study. Patients will be randomly assigned to one of two groups as part of follow-up management: (i) Oral Transmucosal Haloperidol or (ii) Oral Transmucosal Olanzapine.

After commencement of the first dose of medication, each patient will be observed by their family caregiver and the attending clinician over 72 hours (less if the patient dies earlier). Time-points for data collection will be at 24 hours, 48 hours, and 72 hours after first commencement of medication.

This study compares two common treatments in clinical practice, both of which have demonstrated efficacy greater than placebo. Since all participants will receive treatment that is no different from accepted practice, a placebo group was deemed unnecessary and unethical, thus it was not included.

Proxy consent is a method for collecting informed consent, where the proxy (or person responsible) for the potential participant is approached to provide consent on behalf of the prospective participant. Proxy consent was suggested as a suitable method for consent collection, given the patient's absent or fluctuating capacity to consent. It was successfully used in dementia and delirium research, and was reported to have been acceptable to patients and their caregivers.

The clinical staff of the hospice service will be briefed about the study and will assist in recruitment. As they provide standard palliative care to the patient, the clinical staff will (i) identify patients who meet inclusion criteria and share preliminary information with caregivers, (ii) confirm the diagnosis of delirium, and (iii) advise caregivers on appropriate non-pharmacological management.

The primary caregiver (i.e. proxy) will be approached by a study team member who is independent from the management of the patient. They will provide more detailed information about the study to the primary caregiver. If agreeable, the proxy will sign the informed consent form and the dyad is assigned a participant ID number. Basic demographic information, including patient's age, sex, primary diagnosis and co-morbidities will be collected.

Patients may withdraw from the study anytime, without compromising further treatment using other drugs or alternative dosage regimen.

Randomization sequence is created using Microsoft Excel 2016 with 1:1 allocation using random block sizes of 2 and 4. As each participant joins, they are dispensed either haloperidol or olanzapine according to the generated randomization list.

After obtaining consent, the participant-caregiver pair will be randomized into either the Haloperidol or Olanzapine group. Instructions on how to administer the medication will be provided. Caregivers will be advised to serve breakthrough doses of the assigned anti-psychotic drug as needed.

A daily pack of medication will be prepared for the caregiver during daily clinical reviews at home. The pack will have the correct dosages of medication prepared. Subcutaneous (SC) Midazolam is prepared as rescue medication in the event delirium symptoms remain uncontrolled and distressing after the trial medication are depleted.

Per clinical practice, the first dose of medication will be given under the supervision of the study team. The caregiver will be instructed how to rate the patient using the RASS and will provide the baseline RASS rating. The study team will assess the patient's baseline symptom severity with the MDAS.

Alongside drug therapy, usual non-pharmacological interventions will be provided to all patients. These interventions include: (i) regularly orientating the patient, (ii) keeping the room bright during the day, (iii) minimizing the use of tubes, catheters, physical restraints or other immobilizing devices, and (iv) minimizing unnecessary disturbances to the patient.

Every six hours, caregivers will chart the patient's agitation using the RASS. Additionally, if breakthrough medication is required, the time of administration will be documented.

To conduct assessments as well as to ensure patient's safety, the study team will make regular home visits to review the patient 24-hours, 48-hours, and 72-hours after first dose. During each review, the study team will document their assessments of patients' symptom severity (MDAS) and observe for adverse events (NCI CTCAE). The researchers will take appropriate action to ensure patient's safety during the trial, up to and including recommending the termination of the trial.

The trial will be conducted for up to 72 hours after recruitment or until patient's death. If the patient completes the trial and survives, the family will continue to receive support from their primary nurse and attending physician. Patients who survive beyond seven days after recruitment will be excluded from per-protocol analysis, as they no longer fit the inclusion criteria for the study.

The study may be terminated at any point during the trial. In that event, the caregivers will cease assessment using the RASS, while the clinicians will record the reason for cessation, and make a final MDAS and NCI CTC assessment, where applicable. The family will continue to receive support from their primary nurse and attending physician.

The proxy may choose to decline from having the patient participate in the trial. They may also choose to withdraw the patient from the study at any point during the trial. The patient and the family will continue to receive service support from their primary nurse and attending physician thereafter. They will advise how persisting symptoms should be managed, outside of the study. The study team will assure the proxy of this fact before informed consent is collected.

SC Midazolam is prepared as rescue medication in the event the symptoms of delirium remain uncontrolled and distressing. Rescue medications will be used in any one of the following situations:

1. Within 24 hours, the total doses for Haloperidol or Olanzapine reach more than 10mg or 20mg respectively and patient remains unsettled (i.e. all prepared medication are finished any time before the next clinical review).
2. Patient is unable to tolerate Oral Transmucosal medication.
3. Patient experiences serious adverse effects from trial medication.

The study will be terminated for that patient in any one of the following situations:

1. Rescue medication is used.
2. Adverse events related to the trial medication were observed to be intolerable.
3. Caregiver asks to withdraw the patient from the study.
4. Patient is admitted to hospital.

Changes to the severity of delirium are analysed with scores from MDAS. Repeated-measures, between-factors ANOVA will be employed to analyse differences in MDAS scores over time.

If a statistically significant difference is found between medications, post-hoc analysis will be conducted to analyse the change in MDAS scores at each time-point.

Changes in the patient's agitation will be trended using the RASS score. The RASS scores from Baseline, 6 hours, 12 hours, and 24 hours will be analysed. Moreover, an average of the RASS scores for the second day and the third day will be calculated and trended.

Secondary outcomes are possible adverse effects due to the medication, which is measured using NCI CTCAE. For each group, the toxicities (Akathasia, Extrapyramidal disorder, and spasticity) for each group will be compared.

Based on validation studies by Breitbart et al. (1997) and Lawlor et al. (2000), the mean MDAS scores for patients with delirium is roughly 18 (SD = 7.64). Jain et al. (2018) reported that using either Haloperidol or Olanzapine led to nearly 55% reduction in patients' MDAS score (7-8 points). 2 points was estimated to be the minimal important difference between Haloperidol and Olanzapine.

Assuming a data collection period of 27 months and a target recruitment size of 80 participants, the study must successfully recruit 3 - 4 participants per month.

A review of HCA Hospice Care's medical notes from January 2020 to August 2020 found that 250 patients exhibited symptoms of confusion, agitation, or delirium while in an unstable or deteriorating state (approximately 30 patients per month). The duration between the date of these case notes and the date of patient's death ranged 0 days to 17 days; 187 patients died within 7 days. Hence, an average of 23 potential patients per month would be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is above 21 years of age.
2. Patient was diagnosed with a terminal illness and is receiving end-of-life care at home.
3. Patient is assessed to be acutely dying (estimated prognosis of three days or less).
4. Patient is diagnosed with delirium, as described in the DSM-V (American Psychiatric Association, 2013)

Exclusion Criteria:

1. Patient does not have a caregiver at home.
2. Patient has a prior history of dementia, psychosis, schizophrenia or any other mental health issue followed up by psychiatrists or other specialists.
3. Patient is currently receiving, or has been administered Haloperidol or Olanzapine less than a week before participating in the study.
4. Patient has known allergies or adverse reactions to Haloperidol or Olanzapine.
5. Patients who survive 7 days after recruitment will be excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Severity of agitation, measured by the Memorial Delirium Assessment Scale (MDAS) | 72 hours
  MDAS is a ten-item, four-point clinician-rated scale designed to quantify the severity of delirium in medically-ill patients (range 1 - 40). Items included in the scale reflect the diagnostic criteria for delirium in the DSM-IV. It has very good psychometric proper-ties, with high reliability (r = .91) and good Discriminant and Concurrent validity. Though the scale was intended to assess patients based on all ten items, it was suggested that items in MDAS can be pro-rated in the event the patient is not able to communicate.
  The higher the score, the more severe the agitation.
Severity of terminal delirium, measured by the Richmond Agitation-Sedation Scale modified for palliative care (RASS-PAL) | 72 hours
  The RASS is a simple observational instrument assessing levels of sedation and agitation. It requires no patient input and ranges from +4 (overly combative) to -5 (unarousable). It is considered less time-consuming and easier to use than other similar instruments. Developed for adult intensive care unit patients, the scale demonstrated strong inter-rater reliability in that setting. A modified version was de-signed for use in the palliative care setting, which produced acceptable psychometric properties. Hui et. al. (2018) had caregivers using the RASS to assess patients, which gave ratings similar to clinicians.

SECONDARY OUTCOMES:
Adverse effects or toxicity, measured by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) | 0-72 hours
  Possible side effects of taking either drugs are over sedation and extrapyramidal symptoms; these include akathisia, extrapyramidal disorder, and spasticity. To track these adverse events and their severity, the clinician investigator will providing ratings of observed adverse events using the scale provided by the criteria.
  Each symptom is scored between 0 (No symptom) to 3 (Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Poh Heng Chong, MD, Study Director — HCA Hospice Care
Locations (1):
- HCA Hospice Care, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agar M, Ko DN, Sheehan C, Chapman M, Currow DC. Informed consent in palliative care clinical trials: challenging but possible. J Palliat Med. 2013 May;16(5):485-91. doi: 10.1089/jpm.2012.0422. Epub 2013 Apr 30. PMID 23631612
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders: DSM-V (5th ed.). Arlington: American Psychiatric Association.
- [Background] Bannon L, McGaughey J, Verghis R, Clarke M, McAuley DF, Blackwood B. The effectiveness of non-pharmacological interventions in reducing the incidence and duration of delirium in critically ill patients: a systematic review and meta-analysis. Intensive Care Med. 2019 Jan;45(1):1-12. doi: 10.1007/s00134-018-5452-x. Epub 2018 Nov 30. PMID 30506354
- [Background] Breitbart W, Rosenfeld B, Roth A, Smith MJ, Cohen K, Passik S. The Memorial Delirium Assessment Scale. J Pain Symptom Manage. 1997 Mar;13(3):128-37. doi: 10.1016/s0885-3924(96)00316-8. PMID 9114631
- [Background] Bush SH, Grassau PA, Yarmo MN, Zhang T, Zinkie SJ, Pereira JL. The Richmond Agitation-Sedation Scale modified for palliative care inpatients (RASS-PAL): a pilot study exploring validity and feasibility in clinical practice. BMC Palliat Care. 2014 Mar 31;13(1):17. doi: 10.1186/1472-684X-13-17. PMID 24684942
- [Background] Bush SH, Kanji S, Pereira JL, Davis DHJ, Currow DC, Meagher D, Rabheru K, Wright D, Bruera E, Hartwick M, Gagnon PR, Gagnon B, Breitbart W, Regnier L, Lawlor PG. Treating an established episode of delirium in palliative care: expert opinion and review of the current evidence base with recommendations for future development. J Pain Symptom Manage. 2014 Aug;48(2):231-248. doi: 10.1016/j.jpainsymman.2013.07.018. Epub 2014 Jan 28. PMID 24480529
- [Background] Bush SH, Leonard MM, Agar M, Spiller JA, Hosie A, Wright DK, Meagher DJ, Currow DC, Bruera E, Lawlor PG. End-of-life delirium: issues regarding recognition, optimal management, and the role of sedation in the dying phase. J Pain Symptom Manage. 2014 Aug;48(2):215-30. doi: 10.1016/j.jpainsymman.2014.05.009. Epub 2014 May 28. PMID 24879997
- [Background] Casarett DJ, Inouye SK; American College of Physicians-American Society of Internal Medicine End-of-Life Care Consensus Panel. Diagnosis and management of delirium near the end of life. Ann Intern Med. 2001 Jul 3;135(1):32-40. doi: 10.7326/0003-4819-135-1-200107030-00011. PMID 11434730
- [Background] Finucane AM, Jones L, Leurent B, Sampson EL, Stone P, Tookman A, Candy B. Drug therapy for delirium in terminally ill adults. Cochrane Database Syst Rev. 2020 Jan 21;1(1):CD004770. doi: 10.1002/14651858.CD004770.pub3. PMID 31960954
- [Background] Gagnon P, Allard P, Gagnon B, Merette C, Tardif F. Delirium prevention in terminal cancer: assessment of a multicomponent intervention. Psychooncology. 2012 Feb;21(2):187-94. doi: 10.1002/pon.1881. Epub 2010 Dec 19. PMID 22271539
- [Background] Hui D, Dev R, Bruera E. Neuroleptics in the management of delirium in patients with advanced cancer. Curr Opin Support Palliat Care. 2016 Dec;10(4):316-323. doi: 10.1097/SPC.0000000000000236. PMID 27661210
- [Background] Hui D, Hess K, Dibaj SS, Arthur J, Dev R, Dalal S, Reddy S, Bruera E. The minimal clinically important difference of the Richmond Agitation-Sedation Scale in patients with cancer with agitated delirium. Cancer. 2018 May 15;124(10):2246-2252. doi: 10.1002/cncr.31312. Epub 2018 Feb 22. PMID 29469951
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Lawlor PG, Nekolaichuk C, Gagnon B, Mancini IL, Pereira JL, Bruera ED. Clinical utility, factor analysis, and further validation of the memorial delirium assessment scale in patients with advanced cancer: Assessing delirium in advanced cancer. Cancer. 2000 Jun 15;88(12):2859-67. PMID 10870073
- [Background] Mercadante S, Masedu F, Maltoni M, De Giovanni D, Montanari L, Pittureri C, Berte R, Russo D, Ursini L, Marinangeli F, Aielli F. Symptom expression in advanced cancer patients admitted to hospice or home care with and without delirium. Intern Emerg Med. 2019 Jun;14(4):515-520. doi: 10.1007/s11739-018-1969-9. Epub 2018 Oct 17. PMID 30334235
- [Background] Morita T, Hirai K, Sakaguchi Y, Tsuneto S, Shima Y. Family-perceived distress from delirium-related symptoms of terminally ill cancer patients. Psychosomatics. 2004 Mar-Apr;45(2):107-13. doi: 10.1176/appi.psy.45.2.107. PMID 15016923
- [Background] Reston JT, Schoelles KM. In-facility delirium prevention programs as a patient safety strategy: a systematic review. Ann Intern Med. 2013 Mar 5;158(5 Pt 2):375-80. doi: 10.7326/0003-4819-158-5-201303051-00003. PMID 23460093
- [Background] Sweet L, Adamis D, Meagher DJ, Davis D, Currow DC, Bush SH, Barnes C, Hartwick M, Agar M, Simon J, Breitbart W, MacDonald N, Lawlor PG. Ethical challenges and solutions regarding delirium studies in palliative care. J Pain Symptom Manage. 2014 Aug;48(2):259-71. doi: 10.1016/j.jpainsymman.2013.07.017. Epub 2013 Dec 31. PMID 24388124
- [Result] Jain R, Arun P, Sidana A, Sachdev A. Comparison of efficacy of haloperidol and olanzapine in the treatment of delirium. Indian J Psychiatry. 2017 Oct-Dec;59(4):451-456. doi: 10.4103/psychiatry.IndianJPsychiatry_59_17. PMID 29497187
- [Derived] Lyu XJ, Kan AD, Chong PH, Lin K, Koh YH, Yeo ZZ. An open-label clinical trial of oral transmucosal haloperidol and oral transmucosal olanzapine in the treatment of terminal delirium at home. Trials. 2022 Apr 14;23(1):311. doi: 10.1186/s13063-022-06238-4. PMID 35422053